CLINICAL TRIAL: NCT00919048
Title: Uroflow Measurements in Urogynecology Patients Compared to Healthy Female Volunteers
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Gunhilde Buchsbaum, MD, University of Rochester
Other Study IDs: 25597
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Urogynecology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urodynamic patients: Uroflow studies of patients who underwent urodynamics as part of an incontinence work-up.

SUMMARY:
To compare uroflowmetry measurements of patients undergoing urodynamic testing as part of an incontinence work-up in an urogynecology practice to healthy female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent urodynamics at the urogynecology clinic during the past 12 months
* Voids larger than 50 mls.

Exclusion Criteria:

* History of pelvic organ prolapse, incomplete bladder emptying, and voids less than 50cc.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Urogynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Voiding variables of patients will be compared to those of healthy female volunteers collected from another study.

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States